CLINICAL TRIAL: NCT02709772
Title: Provider Alerts to Reduce Unnecessary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul A. Heidenreich, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHCQICW1
Record Dates: First submitted 2016-03-02; First posted 2016-03-16 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Physician's Role

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Provider Alert (Active Comparator): This arm is the intervention arm. This arm will receive the Electronic Record Alert.
  Interventions: Behavioral: Electronic Record Alert
- No Provider Alert (No Intervention): This arm is the control arm.

INTERVENTIONS:
Behavioral: Electronic Record Alert — Electronic alert within the medical record indicating the ordered test or treatment may be inappropriate. The provider can indicate why the test or treatment is appropriate and complete the order.
  Arms: Provider Alert

SUMMARY:
10 Clinics within Stanford Health Care are randomized to receive or not receive provider alerts for 5 commonly overused tests and treatments.

DETAILED DESCRIPTION:
10 Clinics within Stanford Health Care are randomized to receive or not receive provider alerts for 5 commonly overused tests and treatments.

Thus there will potentially be 50 clinics enrolled across the 5 tests/treatment categories. However, it is expected that some clinics will meet criteria to be one of the 10 clinics in more than test/treatment category. Thus the total number of clinics involved will be between 10 and 50.

These 5 tests / treatments are taken from the Choosing Wisely list. All alerts will be provided using the electronic medical record and will be automated.

ELIGIBILITY:
Inclusion Criteria:

High volume clinics defined as the top 10 clinics in Stanford Health Care based on number of electronic orders.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Number of electronic orders entered per 100 clinic patients. | 6 months
  There are five primary outcomes for the five different alerts. For each alert study the outcome will be orders that would qualify for an alert per 100 patients.

SECONDARY OUTCOMES:
Number of potential electronic alerts divided by the number of electronic orders | 6 months
  There will be five secondary outcomes which will be the alert candidate to order ratio. For both the control and intervention groups we will determine the fraction of orders that qualify for an alert.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho VT, Aikens RC, Tso G, Heidenreich PA, Sharp C, Asch SM, Chen JH, Shah NK. Interruptive Electronic Alerts for Choosing Wisely Recommendations: A Cluster Randomized Controlled Trial. J Am Med Inform Assoc. 2022 Oct 7;29(11):1941-1948. doi: 10.1093/jamia/ocac139. PMID 36018731